CLINICAL TRIAL: NCT01545986
Title: A Comparative Analysis of High Velocity and Standard Low Velocity Exercise Training on Rehabilitation Outcomes Following Total Knee Arthroplasty
Brief Title: A Comparative Analysis of Two Types of Exercise on Outcomes Following Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helen Hayes Hospital (Other)
Responsible Party: Principal Investigator, Marie A. Kardys Kelly, Primary Investigator, Helen Hayes Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-04
Record Dates: First submitted 2012-02-26; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Joint Replacement; Exercise; Power training
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Exercise; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Velocity Exercise (Experimental): The high velocity exercise group performed the concentric contraction phase of resisted exercise in one second or less. This group performed sit to stand exercise, walking, curbs, and stairs as fast as was comfortable without an increased limp. Other exercises were performed at the participant preferred rate.
  Interventions: Behavioral: Exercise
- Low Velocity exercise (Active Comparator): The low velocity exercise group performed the concentric contraction phase of resisted exercise in two seconds. This group performed sit to stand exercise, walking, curbs, stairs, and other exercises at the participant preferred rate.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants attended standardized exercise (ex) sessions twice a week for six weeks for 12 sessions. Group speed differed for concentric contractions, sit to stand ex, walking, curbs, and stairs. The low velocity ex group performed a concentric contraction in two seconds, and high velocity group in one second or less. End range concentric hold, eccentric contraction, repetition (rep) rest and set rest were the same. Open chain ex was performed at 50% of one Repetition Maximum (RM) x 10 reps x one set and then 80% of 1RM x 10 reps x two sets. Curb height and 1RM was assessed at the first, fifth and ninth sessions. Manual stretching, balance ex, sit to stand support, level of aerobic ex, gait training, and functional training were assessed and progressed at any session.
  Other Names: Rehabilitation

SUMMARY:
The purpose of this study was to compare the effects of two exercise programs, using low velocity (LV) and high velocity (HV) contractions, on outcomes of individuals who have undergone total knee arthroplasty (TKA). The experimental hypothesis was that individuals performing HV exercise, compared to LV, would exhibit superior outcomes.

DETAILED DESCRIPTION:
The most effective type of exercise has not been identified for individuals who undergo total knee arthroplasty (TKA). High velocity (HV) exercise when compared to low velocity (LV) exercise produces greater gains in power and certain functional activities in older adults. The use of HV exercise for patients who undergo TKA has not been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60- 89 years of age.
* primary unilateral TKA 10-21 days prior to the outpatient PT evaluation
* received inpatient rehabilitation at Helen Hayes Hospital

Exclusion Criteria:

* Any other lower extremity joint or back pain (not inclusive of recent Total knee arthroplasty) rated greater than four out of ten with weight-bearing
* any other lower extremity joint replacement surgery
* diagnosis of osteoporosis with history of fractures, uncontrolled hypertension, unstable cardiac or pulmonary problems, neurological disease affecting motor control, uncontrolled diabetes
* chest pain or shortness of breath on stair-climbing
* requirement of human assistance to walk in addition to the ambulation device
* inability to follow instructions to perform testing and/or exercise,
* participants who stated that they would not be available to complete 12 exercise sessions
* individual adherence with performance of a home exercise program (HEP) less than five of seven days at the end of the treatment period

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Six Minute Walk Test (6MWT) at six weeks | 6 weeks
  The distance walked in six minutes is measured for the 6MWT. A 150 foot hallway is used for the test. Standardized instructions are read to the participant. The participant is asked to walk as fast as he/she feels comfortable and safe in order to walk far as he/she can during six minutes. Distance is recorded in feet and later is converted to meters.

SECONDARY OUTCOMES:
Gait Abnormality Rating Scale (GARS) | 6 weeks
  The GARS is a rating of gait quality. The participant is videotaped walking 10 meters from front, back, left, and right views. No type of walking aid is allowed. Standardized instructions are read to the participant including that he/she should walk at his/her usual speed. At a later time the videotape is viewed to rate gait on a four point (0-3) Likert type scale. Zero is gait without deviations and 48 is greatest amount of gait deviations.
Change from Baseline in Visual Analogue Scale (VAS) Pain at six weeks | 6 weeks
  The VAS Pain is a 10 cm horizontal line with the words "severe moderate slight" spread out along the whole length. The end points are labeled "Pain as bad as it could be" and "No pain". A pencil is given to the participant to mark his/her answer. Standardized instructions are read to the participant. The test is scored by a number from 0 to 100 as measured in mm along the line with zero being no pain and 100 being pain as bad as it could get.
Change from Baseline in Timed Up and Go Test (TUG) at six weeks | 6 weeks
  The TUG records the time in seconds needed to stand from sitting, walk 3 meters, return, and sit into the chair. A standard chair with armrests is used. Assistive devices are allowed but no physical assistance is given. Standardized instructions are read to the participant. A practice walk through is given. Due to the possibility of fatigue the faster of the two times is recorded.
Gait Velocity | 6 weeks
  The participant walks while being videotaped. Standardized instructions are read to the participant when he/she is told that he/she should walk at his/her usual pace to the end of a 10 meter walkway. A side view is used. The videotape is viewed later for scoring. The acceleration and deceleration time is excluded by recording only the time taken to walk across the central 4 meters. This time and the 4 meter distance are used to calculate velocity in meters per second.
Change from Baseline in Short Form-36 (SF-36) at six weeks | 6 weeks
  The Short Form-36 (SF-36) is a 36 item paper questionnaire which measures general health. Standarized instructions read to the participant prior to him/her filling it out. Scores range from 0-100, with 100 being highest level of physical and mental health.
Change from Baseline in Stair Climb Test at six weeks | 6 weeks
  The time used to climb a flight of 12 steps and descend is recorded. Standardized instructions are read to the participant. Time is recorded in seconds. A practice walk through is given. Due to the possibility of fatigue the faster of the two times is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Marie A. Kelly, DHS, Principal Investigator — Helen Hayes Hospital
Locations (1):
- Helen Hayes Hospital, West Haverstraw, New York, United States